CLINICAL TRIAL: NCT04181268
Title: Roller Coaster Trial: Rotational Atherectomy, Lithotripsy or LasER for the Treatment of CAlcified
Brief Title: ROtational Atherectomy, Lithotripsy or LasER for the Treatment of CAlcified STEnosis
Acronym: ROLLERCOASTR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario La Paz (Other)
Responsible Party: Principal Investigator, Alfonso Jurado, MD, PhD, Principal Investigator, Hospital Universitario La Paz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0001
Record Dates: First submitted 2019-11-20; First posted 2019-11-29 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Rotational Atherectomy (Active Comparator): The procedure is performed by using a Rotablator system, which consists of a spring coil shaft with a burr at the tip. The front edge of the burr is the ablating portion, oval shaped, and covered with fine diamond crystals.
  The rotational atherectomy catheter is introduced into the coronary artery over a dedicated long rotational atherectomy wire, which consists of a monofilament stainless steel 0.09-inch wire.
  The device is connected to a console that houses the turbine that rotates the burr with pressurized nitrogen gas. Typically the rpm is set at 150,000 to 180,000 rpm.
  After the lesion is crossed with the wire, the lesion is crossed with multiple "pecking" movements of the burr, with each run lasting not more than 20 seconds. After successful rotational atherectomy with one or more burrs, the procedure is completed with balloon angioplasty and stent placement. This can be achieved by exchanging the rota wire with a workhorse wire and using standard equipment.
  Interventions: Device: Percutaneous coronary Intervention
- Intravascular Lithotripsy (Active Comparator): The procedure is perforemed with a Coronary intravascular lithotripsy (IVL) System that consists of a generator, a connector cable with a push button to allow manually controlled delivery of electric pulses, and semi-compliant balloon catheter.
  The balloon integrates two radiopaque lithotripsy emitters 6 mm that receive electrical pulses from the generator vaporising the fluid within the balloon and creating a rapidly expanding and collapsing bubble. This bubble can transmit unfocused circumferential pulsatile mechanical energy into the vessel wall, in the form of sonic pressure waves equivalent to approximately 50 atmospheres (atm). The IVL therapy consists on a maximun of 8 runs of 10 pulses (80 pulses). The number of therapies needed per lesion will depend on lesion resistance; however, a mínimum of 20 pulses is recommended.
  Alter IVL, an optional additional post-dilatation with non-compliant balloons, a stent is implanted
  Interventions: Device: Percutaneous coronary Intervention
- Excimer Laser (Active Comparator): Excimer laser is pulsed gas laser that use Xenon chloride (XeCl) as the active medium to generate pulses of short wavelength, high-energy ultraviolet (UV) light.
  Excimer laser tissue ablation is mediated through three distinct mechanisms: photochemical, photo-thermal and photomechanical. UV laser light is absorbed by intra-vascular material and breaks carbon-carbon bonds (photochemical). It elevates the temperature of intra-cellular water, causing cellular rupture and generates a vapor bubble at the catheter tip (photo-thermal). Expansion and implosion of these bubbles disrupts the obstructive intra-vascular material (photomechanical). The laser catheter is advanced slowly over a conventional wire while the therapy is aplied and saline is inffused. After laser, balloon dilatation is usually performed finishing the procedure with stent implantation
  Interventions: Device: Percutaneous coronary Intervention

INTERVENTIONS:
Device: Percutaneous coronary Intervention — Calcified plaque modification during percutaneous coronary intervention

SUMMARY:
Some data exist about the efficacy and safety of rotational atherectomy, intravascular lithotripsy and excimer laser to modify calcified plaques.

However there is no direct randomized comparison between these three tools in this scenario.

The aim of this pilot randomized trial is to compare the safety and efficacy of these three techniques during PCI of moderate to severe calcified lesions.

DETAILED DESCRIPTION:
Some data exist about the efficacy and safety of rotational atherectomy, intravascular lithotripsy and excimer laser to modify calcified plaques.

However there is no direct randomized comparison between these three tools in this scenario.

The aim of this pilot randomized trial is to compare the safety and efficacy of these three techniques during PCI of moderate to severe calcified lesions.

The primary endpoint will be the percentage of stent expansion measured with optical coherence tomography. Between secondary endpoints we will analyze the strategy success (defined as successful stent delivery and expansion with <20% residual stenosis and TIMI 3 flow without crossover or stent failure) and presentation of clinical adverse at 1 year follow-up .

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years.
* Stenosis ≥70% in a coronary artery with a diameter ≥2,5 y ≤4 mm.
* Moderate to severe angiographic calcification
* Stable coronary artery disease or NSTEMI.
* Native coronary vessel or bypass graft.

Exclusion Criteria:

* Knwon allergies to aspirin or P2y12 inhibitors.
* STEMI.
* Cardiogenic shock at the time of PCI.
* Treated lesion in a bifurcation with side branch diameter > 2mm.
* Absence of informed consent.
* Impossibility for 1year follow up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-11-15 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Percentage of stent expansion by optical coherence tomography | At the end of percutaneous coronary intervention
  We will analyze with optical coherence tomography the percentage of stent expansion (defined as the minimal stent area divided by the mean of the proximal and distal reference lumen areas).

SECONDARY OUTCOMES:
Strategy success rate | At the end of percutaneous coronary intervention
  Successful stent delivery and expansion with <20% residual stenosis and TIMI3 flow without crossover or stent failure.
  Successful stent delivery and expansion with <20% residual stenosis and TIMI3 flow without crossover or stent failure.
  Successful stent delivery and expansion with residual stenosis <20% and TIMI 3 without crossover

CONTACTS AND LOCATIONS:
Locations (1):
- La Paz University Hospital, Madrid, Spain